CLINICAL TRIAL: NCT02987088
Title: Phase 1 Clinical Trial of Sodium Nitrite for Out of Hospital Cardiac Arrest
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Francis Kim, Associate Professor, Medicine/Division of Cardiology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 51605-A
Record Dates: First submitted 2016-12-03; First posted 2016-12-08 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Sodium Nitrite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sodium Nitrite

SUMMARY:
The purpose of this study is to determine the optimal dose of sodium nitrate administered during resuscitation to achieve a plasma level of 10 μM by hospital arrival.

Pharmacokinetic modeling from human cardiac arrest studies suggest that a single 25 mg IV dose of sodium nitrite will achieve the optimal (based on preclinical studies) neuroprotective plasma levels of 10 μM. In this phase-1 open-label dose finding study in 100 patients, we will determine whether 25 mg IV administered during resuscitation will achieve plasma nitrite levels of at least 10 μM by hospital arrival. Dose adjustments, either decreasing or increasing, will be made if necessary permitting us to determine the optimal nitrite dose needed to achieve the 10 μM plasma target. Safety data will also be collected

ELIGIBILITY:
Inclusion Criteria:

1. Intravenous access/intraosseous access
2. Cardiac arrest, either VF or non-VF patients receiving ACLS by Seattle Medic One paramedics.
3. Age 18 years or older
4. Comatose

Exclusion Criteria:

1. Traumatic cause of cardiac arrest
2. Prisoner, pregnancy, age less than 18 (special population/vulnerable population)
3. Known DNAR
4. Drowning as cause of arrest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-12; Primary Completion 2017-04-05 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
plasma level of sodium nitrite at hospital arrival | 15-45 minutes after dose has been given

SECONDARY OUTCOMES:
Rate of re-arrest | 15-120 minutes after dose has been given
Need for pressor support before hospital arrival | 15-120 minutes after dose has been given

OTHER OUTCOMES:
blood pressure at hospital arrival | at hospital arrival usually 15-60 minutes after cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Francis Kim, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim F, Dezfulian C, Empey PE, Morrell M, Olsufka M, Scruggs S, Kudenchuk P, May S, Maynard C, Sayre MR, Nichol G. Usefulness of Intravenous Sodium Nitrite During Resuscitation for the Treatment of Out-of-Hospital Cardiac Arrest. Am J Cardiol. 2018 Aug 15;122(4):554-559. doi: 10.1016/j.amjcard.2018.04.060. Epub 2018 Jun 20. PMID 30205886